CLINICAL TRIAL: NCT00754156
Title: A Prospective, Controlled Evaluation of ABRA Abdominal Wall Closure System in Combination With V.A.C. Therapy Compared to V.A.C. Alone in the Management of Open Abdomen
Brief Title: ABRA Abdominal Closure System in Open Abdomen Management
Acronym: ABRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Anna Rockich (Other)
Responsible Party: Sponsor-Investigator, Anna Rockich, Director, General Surgery Clinical Research Program, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-0694-F2L
Record Dates: First submitted 2008-09-16; First posted 2008-09-17 (Estimated); Results first posted 2014-03-18 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2014-02

CONDITIONS: Open Abdomen
Keywords: Closure, Wounds
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 ABRA plus KCI ABThera or KCI VAC (Active Comparator): ABRA Abdominal Wound Closure System in combination with KCI ABThera or KCI VAC
  Interventions: Device: V.A.C. Therapy; Device: KCI ABThera
- KCI V.A.C. Therapy or ABThera Alone (Active Comparator): KCI V.A.C. Therapy ABThera Alone
  Interventions: Device: ABRA Abdominal Closure System; Device: V.A.C. Therapy; Device: KCI ABThera

INTERVENTIONS:
Device: ABRA Abdominal Closure System — ABRA Abdominal Closure System
  Arms: KCI V.A.C. Therapy or ABThera Alone
Device: V.A.C. Therapy — V.A.C. Therapy Alone
Device: KCI ABThera — KCI ABThera

SUMMARY:
For the last 20 to 30 years, damage control laparotomy and decompressive laparotomy have emerged as part of the armamentariums for treatment of complex abdominal trauma, abdominal compartment syndrome, and critically ill surgical patients with profound acidosis. While these advances have saved lives, they have also led to a dramatic increase in patients with open abdominal cavities. Various methods have been employed to offer protection to the viscera and at the same time, encourage gradual closure of the abdominal fascia. Some of the techniques have included the Bogota bag, vacuum pack described by Barker , Wittman patch , and the use of vacuum assisted fascia-closure, including the commercially available system offered by KCI. Overall, the abdominal closure rate is approximately 50% to 90% over an average of 10 days. Unfortunately, there has been no well-designed comparison study available. Some of the best results also require returning to the operating room every 3 to 5 days.

At the University of Kentucky Medical Center, a combination of the vacuum pack dressing described by Barker, the commercially available VAC system (V.A.C.; KCI International, San Antonio, TX) and vicryl mesh closure systems are used. The primary fascial closure rate is approximately 50%. It is not standard practice to take patients to the OR every 3-5 days routinely.

Recently, a new FDA listed system (ABRA by Canica) has been introduced using a progressive tension system as a novel approach to the management of open abdomen. ABRA provides a dynamic reduction of full thickness, severely retracted midline abdominal defects with the goal of maintaining or restoring the primary closure option. This subdermal method uses button anchors and elastomer to gradually pull the wound margins together. Tension can be set and adjusted according to the desired outcome; to stabilize a retracted wound, reduce the wound, close the wound or prevent wound dehiscence (Attachment 1: Company brochure). Currently there is only one published case report of the success of this device. We hope to be the first center to prospectively report a series of patients with open abdomen managed with the new ABRA system. In this study, this system will be used in combination with a standard therapy used in abdominal wound closure at the University of Kentucky Medical Center. This system is called the V.A.C system (V.A.C.; KCI International, San Antonio, Tx). This therapy provides active exudate management and containment, assists in reducing abdominal volume and adds structural stabilization to adipose tissue.

Although no highly powered study has been done to establish data on performance, individual experiences at several institutions have reached fascial closure rates of higher than 70% using the ABRA device. One institution in Las Vegas, Nevada is using the ABRA device in combination with the VAC system and has experienced 100% closure rate to date with 12 patients. The purpose of this study is to collect information about the ABRA system in combination with the VAC technique at the University of Kentucky Medical Center. It is our belief that using this system will improve the fascial closure rate and thereby produce less chance of hernia and reduce long periods of open abdominal wounds. The objective of the study is to evaluate a novel approach for closure of open abdomen utilizing the Canica ABRA system combined with the K.C.I. VAC System to KCI VAC System alone.

ELIGIBILITY:
Inclusion Criteria:

1. ages of 18 and 70
2. patients deemed not a candidate for primary fascial closure at the second laparotomy.

Exclusion Criteria:

1. High risk for imminent death, as determined by the attending surgeon and PI
2. Pre-existing large ventral hernia
3. Significant loss of abdominal wall fascia as a result of trauma or infection
4. Known Crohn's disease
5. Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Chang, M.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who met study criteria were enrolled from January 26, 2009 through December 6, 2010.
Pre-assignment Details: Study candidates were identified following index laparotomy where the abdominal cavity could not be closed primarily. Following informed consent, patients were enrolled if attempts at primary closure were unsuccessful during the second laparotomy.
Groups:
- 1 ABRA Plus KCI Abdominal Wound Vac (V.A.C.) or KCI ABThera: ABRA Abdominal Wound Closure System in combination with ABThera V.A.C. Therapy
- 2 V.A.C. or ABThera Alone: ABThera V.A.C. Therapy alone
Period: Overall Study
Arm/Group | 1 ABRA Plus KCI Abdominal Wound Vac (V.A.C.) or KCI ABThera | 2 V.A.C. or ABThera Alone
Started | 8 | 6
Completed | 8 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1 ABRA Plus V.A.C or ABThera: ABRA Abdominal Wound Closure System in combination with V.A.C. or AbThera Therapy
- V.A.C. or ABThera: V.A.C. or ABThera Therapy alone
- Total: Total of all reporting groups
Arm/Group | 1 ABRA Plus V.A.C or ABThera | V.A.C. or ABThera | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (12.4) | 52.8 (14.1) | 51.14 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 7 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 14
BMI [Mean (Standard Deviation); unit: Kg/m^2] — Body Mass Index
  Kg/m^2 | 25.7 (5.8) | 38.0 (12.9) | 30.99 (2.95)
Base Excess/Base Deficit [Median (Inter-Quartile Range); unit: mmole/liter] — In human physiology, base excess and base deficit refer to an excess or deficit, respectively, in the amount of base present in the blood. The value is usually reported as a concentration in units mmol/L, with a positive number indicating excess of base and a negative deficit. A range for base excess or base deficit is -3 to + 3 mmol/L
  mmole/liter | 5.9 (2.5-18.1) [-4.9 to 19.8] | 5.1 (0.5-9.8) [-2.4 to 15] | 5.9 [-4.9 to 19.8]
APACHE II [Mean (Standard Deviation); unit: score] — APACHE II (Acute Physiology and Chronic Health Evaluation) scoring system is an objective assessment of severity of illness in patients in the ICU. Scores can range from 0 (low severity) to 71 (high severity).
  score | 21.25 (9.8) | 16 (11.6) | 19.00 (2.81)
Starting Wound Dimension [Mean (Standard Deviation); unit: cm^2] | 575.9 (289.2) | 359.2 (245.3) | 483 (75.86)
Trauma [Number; unit: participants] — Number of patients that are trauma patients
  participants | 3 | 2 | 5
Vascular/Splenectomy/AAA [Number; unit: participants] — Patients who met criteria for entry who had baseline conditions to include vascular issue or splenectomy
  participants | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Primary Closure Rate
Description: The rate in which the abdomen was closed the first time.
Time Frame: up to 12 months
Population: Descriptive Study.
Measure: Number; unit: % of participants
Groups:
- 1 ABRA Plus ABThera: ABRA Abdominal Wound Closure System in combination with ABThera V.A.C. Therapy
- 2 ABThera: ABThera V.A.C. Therapy alone
Arm/Group | 1 ABRA Plus ABThera | 2 ABThera
Number analyzed (Participants) | 8 | 6
% of participants | 75 | 67

2. Primary Outcome: Number of Trips to the Operating Room
Time Frame: 12 Months
Measure: Median (Inter-Quartile Range); unit: Number of trips
Groups:
- 1 ABRA Plus ABThera: ABRA Abdominal Wound Closure System in combination with V.A.C or ABThera V.A.C. Therapy
- 2 ABThera: V.A.C. or ABThera V.A.C. Therapy alone
Arm/Group | 1 ABRA Plus ABThera | 2 ABThera
Number analyzed (Participants) | 8 | 6
Number of trips | 1 [1 to 1] | 3 [2.8 to 4.8]

3. Primary Outcome: Operating Room Time Utilization
Description: The amount of time needed to manage the open abdomen inside the operating room.
Time Frame: Duration of Hospital Stay less than 6 months
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- 1 ABRA Plus V.A.C. or ABThera: ABRA Abdominal Wound Closure System in combination with V.A.C. or ABThera V.A.C. Therapy
- 2 V.A.C. or ABThera Alone: V.A.C. or ABThera V.A.C. Therapy alone
Arm/Group | 1 ABRA Plus V.A.C. or ABThera | 2 V.A.C. or ABThera Alone
Number analyzed (Participants) | 8 | 6
Minutes | 58 (29) | 212 (115)
Statistical Analysis 1: Comparison: 1 ABRA Plus V.A.C. or ABThera vs 2 V.A.C. or ABThera Alone; Test type: Non-Inferiority or Equivalence — Equivalence analysis; p < 0.01, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Days to Closure
Time Frame: Duration of Hospital Stay less than 6 months
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | 1 ABRA Plus KCI Abdominal Wound Vac (V.A.C.) or KCI ABThera | 2 V.A.C. or ABThera Alone
Number analyzed (Participants) | 8 | 6
Days | 9.5 [4.5 to 18.0] | 7.5 [5.56 to 10.3]

5. Secondary Outcome: ICU Days
Time Frame: Duration of hospital stay less than 6 months
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | 1 ABRA Plus KCI Abdominal Wound Vac (V.A.C.) or KCI ABThera | 2 V.A.C. or ABThera Alone
Number analyzed (Participants) | 8 | 6
Days | 17 [12.3 to 55.0] | 18 [15.0 to 23.8]

6. Secondary Outcome: Hospital Days
Time Frame: Duration of Hospital Stay less than 6 months
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | 1 ABRA Plus KCI Abdominal Wound Vac (V.A.C.) or KCI ABThera | 2 V.A.C. or ABThera Alone
Number analyzed (Participants) | 8 | 6
Days | 43.5 [22.3 to 60.8] | 27.5 [25.8 to 31.5]

7. Secondary Outcome: Blood Transfused
Time Frame: Duration of Hospital Stay less than 6 months
Measure: Median (Inter-Quartile Range); unit: Units
Arm/Group | 1 ABRA Plus KCI Abdominal Wound Vac (V.A.C.) or KCI ABThera | 2 V.A.C. or ABThera Alone
Number analyzed (Participants) | 8 | 6
Units | 2650 [0 to 7493] | 0 [0 to 758]

ADVERSE EVENTS:
Time Frame: Hospitalization of enrollment
Arm/Group | 1 ABRA Plus KCI Abdominal Wound Vac (V.A.C.) or KCI ABThera | 2 V.A.C. or ABThera Alone
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/6
Other Adverse Events (participants affected / at risk) | 0/8 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 ABRA Plus KCI Abdominal Wound Vac (V.A.C.) or KCI ABThera (N=8) | 2 V.A.C. or ABThera Alone (N=6)
Device failure and skin breakdown (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Mass amount of drainage and infection and absence of wound edge for > 3 days required ABRA removal. Following removal 2 JP drains and wound vac was required. Soft tissue debridement was needed where the ABR button pads rested.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 ABRA Plus KCI Abdominal Wound Vac (V.A.C.) or KCI ABThera (N=8) | 2 V.A.C. or ABThera Alone (N=6)
Enterocutaneous Fistula (Surgical and medical procedures) | 0 (0) | 1 (1) — This patient developed an entercutaneous fistula during her involvement with the study. She recovered without issue

LIMITATIONS AND CAVEATS:
1. Limited by small sample size, and lack of closely matched patient groups.
2. Limited by product change from the original VAC to the ABThera system mid study.
3. Limited by a significant learning curve in application and use of the ABRA device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other